CLINICAL TRIAL: NCT06913075
Title: Is GnRH Agonist Plus Letrozole a Better Choice Than GnRH Agonist Alone in Adenomyosis Cases Undergoing Frozen Embryo Transfer?
Brief Title: FET in Adenomyosis
Acronym: ADY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indira IVF Hospital Pvt Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIHL/UDR/P/003_2024
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Adenomyosis
Keywords: Frozen embryo transfer; Adenomyosis; ongoing pregnancy rate; live birth rate
MeSH Terms: conditions — Adenomyosis | interventions — Gonadotropin-Releasing Hormone; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Drug: GnRH agonist downregulation
- Group B (Active Comparator)
  Interventions: Drug: GnRH agonist and Letrozole

INTERVENTIONS:
Drug: GnRH agonist downregulation — Triptorelin Acetate 3.75mg for two consecutive dosage at 30 days interval
  Arms: Group A
Drug: GnRH agonist and Letrozole — Triptorelin Acetate 3.75mg for two consecutive dosages at 30 days interval) + Letrozole (5 mg once daily for a total of 21 days during the second depot - letrozole stops when Estrogen priming starts
  Arms: Group B

SUMMARY:
Purpose of the Study:

To compare the effectiveness of GnRH agonist downregulation alone versus GnRH agonist combined with letrozole in improving pregnancy outcomes in women with adenomyosis undergoing frozen embryo transfer (FET).

Research Question:

Is the combined use of GnRH agonist and letrozole more effective than GnRH agonist downregulation alone in achieving better ongoing pregnancy rates in adenomyosis cases undergoing FET?

Hypothesis:

Null Hypothesis (H₀): The combined use of GnRH agonist and letrozole is not more effective than GnRH agonist downregulation alone in achieving a higher ongoing pregnancy rate in adenomyosis cases undergoing FET.

Study Outcomes:

Primary Outcome: Ongoing pregnancy rate at 12 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of adenomyosis confirmed via transvaginal ultrasound as per MUSA criteria History of infertility requiring frozen embryo transfer (FET). Availability of at least one good-quality frozen embryo for transfer

Exclusion Criteria:

BMI ≥ 30 kg/m2 Presence of endocrine disorders; (uncontrolled diabetes mellitus, / hyperprolactinemia, thyroid dysfunction, Congenital adrenal hyperplasia, Cushing syndrome, or polycystic ovary syndrome Previous major uterine surgery Gestational carrier Fertility preservation

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with adenomyosis who are undergoing frozen embryo transfer (FET) as part of their fertility treatment.
Enrollment: 700 (Estimated)
Dates: Start 2026-06-25 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks of gestation
  Presence of gestational sacs with a heartbeat at the 12th gestational week. The ongoing pregnancy rate will be calculated using the below formula.
  Ongoing pregnancy rate: (the number of ongoing pregnancy cases/the number of clinical pregnancy cases) × 100%

SECONDARY OUTCOMES:
Implantation Rate | 4 weeks after embryo transfer
  The number of gestational sacs observed by transvaginal ultrasound at the 6th gestational week per the number of embryos transferred. The implantation rate will be calculated using the below formula.
  Implantation rate: (The number of gestational sacs observed/ number of embryos transferred) × 100
Chemical Pregnancy rate | 4 weeks after embryo transfer
  Detection of a fetal heartbeat on transvaginal ultrasound at the 6th gestational week. The clinical pregnancy rate will be calculated using the below formula.
Biochemical loss rate | 4 weeks after embryo transfer
  Pregnancies diagnosed only by β-human chorionic gonadotropin detection without a gestational sac visualized by vaginal ultrasound at the 6th gestational week. The biochemical loss rate will be calculated using the below formula.
  Biochemical loss rate: (the number of biochemical pregnancy loss cases/the number of women per group) × 100%
1st trimester loss | 12 weeks of gestation
  First-trimester loss refers to the spontaneous loss of a pregnancy occurring before the end of the 12th week of gestation
2nd trimester loss | 20 weeks of gestation
  Second-trimester loss refers to the spontaneous loss of a pregnancy occurring between 13 and 20 weeks of gestation.
Live Birth Rate | Post delivery after completion of 20 weeks of gestation
  The number of deliveries that resulted in at least one live birth per 100 Embryo transferred cycle.
  Live birth rate: (The number of live births / the number of embryos transferred cycle) × 100

CONTACTS AND LOCATIONS:
Locations (1):
- Indira IVF Pvt Hospital, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Yes
he Individual Participant Data (IPD) will be shared with authorized researchers upon request. The supporting documents, including the study protocol, SAP, and ICF, will be provided alongside the IPD to ensure comprehensive understanding and proper data interpretation.
  When: IPD will be available after the completion of the study and publication of primary results.
  How: IPD will be shared through a secure data repository or via encrypted files sent through secure email upon request, following proper data use agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication

REFERENCES:
- [Result] Salim R, Riris S, Saab W, Abramov B, Khadum I, Serhal P. Adenomyosis reduces pregnancy rates in infertile women undergoing IVF. Reprod Biomed Online. 2012 Sep;25(3):273-7. doi: 10.1016/j.rbmo.2012.05.003. Epub 2012 May 23. PMID 22832421
- [Result] Younes G, Tulandi T. Effects of adenomyosis on in vitro fertilization treatment outcomes: a meta-analysis. Fertil Steril. 2017 Sep;108(3):483-490.e3. doi: 10.1016/j.fertnstert.2017.06.025. PMID 28865548
- [Result] Han B, Liang T, Zhang W, Ma C, Qiao J. The effect of adenomyosis types on clinical outcomes of IVF embryo transfer after ultra-long GnRH agonist protocol. Reprod Biomed Online. 2023 Feb;46(2):346-351. doi: 10.1016/j.rbmo.2022.09.021. Epub 2022 Sep 26. PMID 36549997
- [Result] Sharma S, RoyChoudhury S, Bhattacharya MP, Hazra S, Majhi AK, Oswal KC, Chattopadhyay R. Low-dose letrozole - an effective option for women with symptomatic adenomyosis awaiting IVF: a pilot randomized controlled trial. Reprod Biomed Online. 2023 Jul;47(1):84-93. doi: 10.1016/j.rbmo.2023.03.010. Epub 2023 Mar 18. PMID 37149412
- [Result] Li Y, Ge L, Yang X, Cui L, Chen ZJ. Effects of duration of long-acting GnRH agonist downregulation on assisted reproductive technology outcomes in patients with adenomyosis: a retrospective cohort study. Front Med (Lausanne). 2023 Sep 26;10:1248274. doi: 10.3389/fmed.2023.1248274. eCollection 2023. PMID 37822471